CLINICAL TRIAL: NCT07073248
Title: Neuroplastic Changes and Effects of Intermittent Theta Burst Stimulation (iTBS) on Motor Recovery of Upper and Lower Extremity in Chronic Stroke Patients
Brief Title: Effects of Intermitted Theta Burst Stimulation (iTBS) on Motor Recovery of Upper Extremity in Chronic Stroke Patients
Acronym: NIMBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Associate Professor, Reg Physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: iTBS-study upper extremity
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemiplegia; Hemiparesis After Stroke; Hand Functionality; Chronic Stroke Patients
Keywords: stroke; iTBS; TMS; Motor cortex; chronic stroke patients; hand dexterity; Hemiparesis; Transcrania Magnetic Stimulation; intermittent Theta Burst Stimulation
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipsilesional motor cortex iTBS and conventional rehabilitation (Experimental): The experimental group will receive intermittent theta burst stimulation on the ipsilesional motor cortex followed by 45 minutes of conventional rehabilitation interventions involving the upper extremity led or instructed by a physiotherapist.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Ipsilesional motor cortex sham-iTBS and conventional rehabilitation (Sham Comparator): The placebo group will receive sham intermittent theta burst stimulation on the ipsilesional motor cortex followed by 45 minutes of conventional rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist.
  Interventions: Device: Sham Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — iTBS protocol: 600 pulses at 80% of AMT for 190 sec on the ipsilesional motor cortex, targeted with the support of a neuronavigational system, 15 sessions over a period of 5 weeks
  Other Names: iTBS; TMS
  Arms: Ipsilesional motor cortex iTBS and conventional rehabilitation
Device: Sham Intermittent Theta Burst Stimulation — It is identical to its active version, replicates operational sounds, and delivers a very shallow magnetic field to mimic the sensation of magnetic stimulation
  Arms: Ipsilesional motor cortex sham-iTBS and conventional rehabilitation

SUMMARY:
This study aims to evaluate the effects and clinical feasibility of non-invasive brain stimulation protocols, specifically intermittent Theta Burst Stimulation, as part of rehabilitation interventions for motor recovery of upper extremity in the chronic phase after stroke.

It also seeks to explore the underlying mechanisms by investigating changes of functional and structural brain networks.

DETAILED DESCRIPTION:
In this randomized controlled trial (RCT) group A will receive iTBS while group B will receive sham iTBS. Both groups will directly after the intervention receive 45 minutes of conventional physical therapy 3 times per week for 5 weeks, a total of 15 interventions by a blinded physiotherapist. For the iTBS intervention a Magstim Rapid² stimulator will be used also equipped with a Cadwell Sierra Summit EMG system [for motor evoked potential (MEP) measurements] and an ANT Visor2™ neuronavigation system [for navigated transcranial magnetic stimulation (TMS) interventions]. The iTBS parameters that will be used are: 600 pulses under 190 seconds at 80 % of Active Motor Threshold (AMT). The ipsilesional motor cortex will be targeted. The participants and clinical assessors will be blinded to the intervention.

All the patients will undergo advanced neuroimaging examinations before and after the intervention period. The exams will be then compared to identify neuroplastic changes in brain circuits.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Chronic stroke (>6 months)
* Residual hemiparesis FM-UE>17

Exclusion Criteria:

* Metal implants
* Epilepsy/seizures
* Pregnancy
* Claustrophobia (related to MRIs exams)
* Severe cognitive impairment
* Untreated or unstable depression/anxiety
* Other disabilities prohibiting intensive physical training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  used to quantify recovery of sensorimotor function in the upper extremity after a stroke. It is a 63 item test scored on a 3-level ordinal scale. The score ranges from 0 to 126 points. A higher score indicates recovery of sensorimotor function.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Assesses spasticity on a 6 point scale/muscle (0p no impairment, 5p max impairment/muscle)
Neuroflexor | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Medical technology device. Assesses spasticity by identifying the neural, viscous and elastic components during passive movement using a biomechanical algorithm (presented in Newton)
Box and Block Test (BBT) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  measures unilateral gross manual dexterity. The score is based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Higher scores indicate better manual dexterity.
Action Research Arm Test (ARAT) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  assesses upper extremity activity capacity in people with stroke. It is a 19-item test scored on a 4-level ordinal scale (0-3). The score ranges from 0 to 57. Higher scores indicate better performance of the upper extremity.
Dextrain Manipulandum™ | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  allows measurement of flexion-extension finger movements. Force sensors are incorporated in the ergonomically designed tool allowing precision measurement of finger movements. The tool is coupled with specific exercises for evaluation of key components of manual dexterity.
Hand-held Dynamometer/Grip Strength | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  A quantitative and objective measure of isometric muscular strength of the hand and forearm. This instrument is scored using force production: kilograms or pounds. Maximum grip is the mean of three trials.
Purdue Pegboard Test (PPT) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  is a test of fingertip dexterity and gross movement of the hand, fingers and arm in patients with impairments of the upper extremity resulting from neurological and musculoskeletal conditions. Number of correctly placed pinns within a time frame are counted and a higher scores indicate better dexterity.
Visuomotor force tracking | At baseline and after completion of the 5 week intervention and at the 12 weeks follow up, to assess changes
  Subjects perform a visually guided, isometric precision grip ramp-and-hold force-tracking task by holding a manipulandum. The standardized visuomotor ramp-and-hold task is performed by following the target force with a cursor on a screen as precisely as possible.
Montreal Cognitive Assessment (MoCA) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Assesses mental function (0p max impairment summed up to 30p no detected impairment)
Canadian Occupational Performance Measure | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Capture the participant´s perception of performance in everyday living and will be used to set goals for the intervention.
Stroke Impact Scale (SIS) | At baseline and after completion of the 5 week intervention and at the 12 weeks follow up, to assess changes
  is a self-report questionnaire that evaluates disability and health-related quality of life after stroke. It has 8 domains: strength, hand function, mobility, physical and instrumental activities of daily living (ADL and IADL), memory and thinking, communication, emotion, and social participation. It uses a 5-point Likert scale to assess the difficulty of performing various tasks within each domain. Higher scores indicate better outcome.
Motor Evoked Potentials (MEPs) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  electrical signals recorded from neural tissue or muscle following activation of central motor pathways. MEPs assess the integrity of descending motor pathways.
Resting state functional MRI (rs-fMRI) | At baseline and after completion of the 5 week intervention to assess changes.
  a method aimed at examining intrinsic networks in the brain while no task is performed (rest); this is to estimate correlations between brain regions.
Diffusion Tension Imaging (DTI) | At baseline and after completion of the 5 week intervention to assess changes.
  a method aimed at mapping structural correlations between brain regions.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | At baseline
  quantifies stroke severity based on weighted evaluation findings. The total NIHSS score ranges from 0 to 42, with higher scores indicating more severe strokes, categorized as follows: minor stroke (1-4), moderate stroke (5-15), moderate to severe stroke (16-20), and severe stroke (21-42).
Barthel Index (BI) | At baseline.
  measures a person's ability to complete activities of daily living (ADL). Scores range from 0 to 100, categorized as follows: Total dependence (0-20), Severe dependence (21-60), Moderate dependence (61-90), Slight dependence (91-99), and Independence (100).
Theoretical Framework of Acceptability questionnaire | After completion of the 5 week intervention to assess acceptability.
  to assess the acceptability of healthcare interventions, based on the developed Theoretical Framework of Acceptability (TFA). It uses a 5-point Likert scale to assess acceptability of the intervention. Higher scores indicate higher acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Palmcrantz, PhD, Associate Professor, Principal Investigator — Dep of Clinical Sciences, Karolinska Institutet
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm 18288, Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemon RN. Descending pathways in motor control. Annu Rev Neurosci. 2008;31:195-218. doi: 10.1146/annurev.neuro.31.060407.125547. PMID 18558853
- [Background] Zhang JJ, Bai Z, Fong KNK. Priming Intermittent Theta Burst Stimulation for Hemiparetic Upper Limb After Stroke: A Randomized Controlled Trial. Stroke. 2022 Jul;53(7):2171-2181. doi: 10.1161/STROKEAHA.121.037870. Epub 2022 Mar 23. PMID 35317611
- [Background] Zhang JJ, Sui Y, Sack AT, Bai Z, Kwong PWH, Sanchez Vidana DI, Xiong L, Fong KNK. Theta burst stimulation for enhancing upper extremity motor functions after stroke: a systematic review of clinical and mechanistic evidence. Rev Neurosci. 2024 Apr 29;35(6):679-695. doi: 10.1515/revneuro-2024-0030. Print 2024 Aug 27. PMID 38671584
- [Background] Jiang T, Wei X, Wang M, Xu J, Xia N, Lu M. Theta burst stimulation: what role does it play in stroke rehabilitation? A systematic review of the existing evidence. BMC Neurol. 2024 Feb 1;24(1):52. doi: 10.1186/s12883-023-03492-0. PMID 38297193
- [Background] van Lieshout ECC, van der Worp HB, Visser-Meily JMA, Dijkhuizen RM. Timing of Repetitive Transcranial Magnetic Stimulation Onset for Upper Limb Function After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2019 Dec 3;10:1269. doi: 10.3389/fneur.2019.01269. eCollection 2019. PMID 31849827
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Christiansen MG, Senko AW, Anikeeva P. Magnetic Strategies for Nervous System Control. Annu Rev Neurosci. 2019 Jul 8;42:271-293. doi: 10.1146/annurev-neuro-070918-050241. Epub 2019 Apr 2. PMID 30939100
- [Background] Fan H, Song Y, Cen X, Yu P, Biro I, Gu Y. The Effect of Repetitive Transcranial Magnetic Stimulation on Lower-Limb Motor Ability in Stroke Patients: A Systematic Review. Front Hum Neurosci. 2021 Sep 1;15:620573. doi: 10.3389/fnhum.2021.620573. eCollection 2021. PMID 34539362